CLINICAL TRIAL: NCT00519389
Title: A Phase I/IIa Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of an H5N1 Virus-Like Particle (VLP) Influenza Vaccine (Recombinant)
Brief Title: Safety, Reactogenicity and Immunogenicity of an H5N1 VLP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H5N1 VLP-1
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2012-03

CONDITIONS: Pandemic Influenza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose H5N1 VLP Vaccine (Experimental)
  Interventions: Biological: H5N1 VLP Vaccine
- Mid dose H5N1 VLP Vaccine (Experimental)
  Interventions: Biological: H5N1 VLP Vaccine
- High dose H5N1 VLP Vaccine (Experimental)
  Interventions: Biological: H5N1 VLP Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: H5N1 VLP Vaccine — Two doses - Day 0 & Day 28
  Arms: High dose H5N1 VLP Vaccine; Low dose H5N1 VLP Vaccine; Mid dose H5N1 VLP Vaccine
Biological: Placebo — Two doses - Day 0 & Day 28
  Arms: Placebo

SUMMARY:
This is a Phase I/IIa randomized, double-blind, placebo-controlled study to evaluate the safety, reactogenicity, and immunogenicity of 3 potencies (dosages) of H5N1 VLP vaccine or placebo in healthy adults 18 to 40 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 40 years of age at the time of the vaccination.
2. Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., return for follow-up visits and completion of the data collection tool).
3. Available by telephone.
4. Free of obvious health problems as established by medical history and clinical examination before entering the study.
5. If subject is of childbearing potential, she must be abstinent or have used adequate contraceptive precautions (e.g., intrauterine contraceptive device; oral contraceptives or other equivalent hormonal contraception) for 30 days prior to vaccination. She must also have a negative pregnancy test at study entry and must agree to continue such precautions for two months after completion of vaccination.
6. Must provide written, informed consent.

Exclusion Criteria:

1. Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
2. Has received any other licensed vaccines within 4 weeks prior to enrollment in this study.
3. Has received any influenza vaccine within the prior 12 month period.
4. Has received any investigational vaccine designed for protection against avian influenza.
5. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine. The use of inhaled and nasal steroids will be permitted.
6. Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
7. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or during the study.
8. Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever ≥ 100.5º F.
9. Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
10. Major congenital defects or serious chronic illness.
11. History of any neurological disorders or seizures, with the exception of febrile seizures during childhood.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety and reactogenicity of H5N1 VLP Vaccine | 6 months

SECONDARY OUTCOMES:
Immunogenicity of H5N1 VLP Influenza vaccine | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: George Atiee, M.D., Principal Investigator — Healthcare Discoveries, Inc.
Locations (1):
- Healthcare Discoveries, Inc., San Antonio, Texas, United States